CLINICAL TRIAL: NCT02449408
Title: Novel Screening Tools For the Evaluation and Management of Malnourished Children in the Developing World
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00058058
Record Dates: First submitted 2015-05-18; First posted 2015-05-20 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Overweight, Obesity, Small for Gestational Age, Prematurity
MeSH Terms: conditions — Overweight; Obesity; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Overweight or Obese: Children being seen in consultation or follow-up within the Duke Division of Pediatric Endocrinology and Diabetes who are overweight or obese.
  Interventions: Other: Measurement of leptin and adiponectin obtained through blood sampling via venipuncture or finger/heelstick using novel screening tool
- Premature or Small for Gestational Age: Infants hospitalized in the Duke Transitional Care Nursery who were born prematurely or small for gestational age.
  Interventions: Other: Measurement of leptin and adiponectin obtained through blood sampling via venipuncture or finger/heelstick using novel screening tool

INTERVENTIONS:
Other: Measurement of leptin and adiponectin obtained through blood sampling via venipuncture or finger/heelstick using novel screening tool

SUMMARY:
The purpose of this study is to evaluate the accuracy of a new device that may be used for the evaluation and management of malnourished infants and children. The device will measure the levels of two hormones made by fat tissue: leptin and adiponectin.

DETAILED DESCRIPTION:
The purpose of this study is to validate novel screening tools for the evaluation and management of malnourished infants and children in the developing world. The study will validate 2-D diffusion point of care testing (POCT) for the rapid analysis of leptin and adiponectin, as these cytokines have been shown to predict mortality in malnourished infants and children. The study will enroll 20 participants, 10 overweight or obese adolescents presenting to the Duke Division of Pediatric Endocrinology outpatient clinics, in whom leptin is expected to be high and adiponectin low, and 10 premature or small for gestational age infants hospitalized in the Duke Transitional Care Nursery, in whom leptin is expected to be low and adiponectin high. Informed consent will be obtained and 0-1 mL of blood will be collected and analyzed using the 2-D POCT and commercial ELISA assays. To reduce potential risks associated with venipuncture and/or finger or heelstick, blood draws for the purposes of this study will take place only when blood sampling is performed at the request of the primary provider, and an attempt will be made to utilize scavenge samples from infants where applicable. The POCT will be validated against the commercial ELISA assays. The investigators will analyze the results of each assay in addition to the means and standard deviations of the POCT and ELISAs and will consider the POCT valid if their variation from ELISA is <20%. The long-term goal of this project is to utilize this novel technology to identify and treat high-risk malnourished infants and children before they have reached the stage of critical, life-threatening illness.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or Obese: Inclusion criteria for these subjects will include:

  1. Age 8-17 years;
  2. male or female; and
  3. BMI >85% for age.
* Premature or Small for Gestational Age: Inclusion criteria for these subjects will include:

  1. Age <1 year,
  2. male or female,
  3. small for gestational age or intra-uterine growth restriction (IUGR) defined by the 9th revision of the International Classification for Diseases OR
  4. prematurity as defined by the 9th revision of the International Classification for Diseases.

Exclusion Criteria:

* Exclusion criteria include refusal or inability to provide samples of blood.

Ages: 1 Hour to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The investigators plan to recruit 10 overweight or obese adolescents followed by the Duke Division of Pediatric Endocrinology and Diabetes. Investigators will review the electronic medical records of potential participants identified by their primary providers to ensure they meet the eligibility criteria.
  The investigators will also recruit 10 infants hospitalized in the Duke Transitional Care Nursery and will review the electronic medical records of potential participants identified by their primary providers to ensure they meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Variation between results of novel screening tool and standard ELISA | 1 year
  The 2-D diffusion POCT will be validated against commercial ELISA assays, run in the Duke Molecular Physiology Institute laboratory, using recombinant human leptin and high molecular weight adiponectin from blood samples. Dose-response curves will be generated using analyte-spiked buffer. The dose-response data from 20 separate dose-response dilutions will be fit with the five-parameter logistic (5-PL) curve. The coefficients of variation (inter and intra-assay) for standard ELISAs for leptin and adiponectin assays are less than 10%. The investigators will analyze the results of each assay in addition to the means and standard deviations of the POCT assays and ELISAs. The POCT assay will be considered valid if the variation from the ELISA is less than 20% and if there is no statistically significant difference between the means and standard deviations.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States